CLINICAL TRIAL: NCT05972941
Title: The Effect of Nicotine and Tobacco Message Framing on Use Among Diverse Groups of Young Adults
Brief Title: Nicotine and Tobacco Message Framing Among LGBT Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joanne Patterson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OSU-23020; 4R00CA260718-02 (NIH); NCI-2024-05891 (Other: NCI)
Record Dates: First submitted 2023-06-26; First posted 2023-08-02 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Tobacco-Related Carcinoma
Keywords: health communication; LGBT
MeSH Terms: interventions — Health Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally targeted messages (Experimental): Participants will view 8 nicotine and tobacco health messages with LGBT culturally targeted messages and imagery
  Interventions: Behavioral: Health communications
- Non-targeted messages (Other): Participants will view 8 nicotine and tobacco health messages with universal messages and imagery
  Interventions: Behavioral: Health communications

INTERVENTIONS:
Behavioral: Health communications — Participants will view eight culturally targeted or non-targeted health communications about the health risks of nicotine and tobacco use.

SUMMARY:
This trial refines and evaluates how cultural targeting influences the effectiveness of anti-tobacco messages among lesbian, gay, bisexual, and transgender (LGBT) young adults at risk for the use of more than one tobacco product (polytobacco use). Polytobacco use is associated with nicotine dependence and tobacco use into adulthood, and is disproportionately high among LGBT young adults. This trial seeks to determine how cultural targeting can be applied to communicate polytobacco use risk to at-risk LGBT young adults.

DETAILED DESCRIPTION:
The goal of this study is to identify if culturally targeted (CT) or non-targeted (NT) anti-polytobacco messages are most effective for engaging LGBT consumers. Using the most effective NT messages from Aim 1, investigators will create a set of CT messages. Message framing will remain consistent between CT and NT messages; however, CT messages will include language and graphics representing LGBT values formative research and the existing peer-reviewed literature. Participants will be randomized to view CT or NT messages in a virtual lab where investigators will assess eye-tracking, self-reported perceived effectiveness, risk perceptions, and behavioral intentions. Participants will also complete a 1-week follow-up. The study aims to determine the effects of cultural targeting on attention to anti-polytobacco messages and perceived effectiveness among LGBT young adults susceptible to polytobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English fluently
* Self-identifies as lesbian, gay, bisexual, transgender, queer, or another non- heterosexual orientation or non-binary gender identity
* Ever used e-cigarettes AND combustible cigarettes
* Currently uses e-cigarettes, combustible cigarettes, or both e-cigarettes and combustible cigarettes
* Resides in the United States
* Access to a laptop or desktop computer with a camera for virtual eye-tracking

Exclusion Criteria:

* Glaucoma
* Cataracts

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne G Patterson, PhD, Principal Investigator — The Ohio State University College of Public Health
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who consented to the study but did not complete the activity in REDCap that triggered randomization to an arm, were excluded from the rest of the study.
Groups:
- Culturally Targeted Messages: Participants will view 8 nicotine and tobacco health messages with lesbian, gay, bisexual, and transgender (LGBT) culturally targeted messages and imagery
Period: Overall Study
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Started | 129 | 122
Completed | 83 | 82
Not Completed | 46 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Culturally Targeted Messages | Non-targeted Messages | Total
Number analyzed (Participants) | 129 | 122 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 129 | 122 | 251
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 61 | 64 | 125
  Male | 44 | 33 | 77
  Unknown | 24 | 25 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 11 | 15
  Not Hispanic or Latino | 123 | 110 | 233
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 17 | 11 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 54 | 59 | 113
  White | 52 | 49 | 101
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 129 | 122 | 251
Behavioral Intentions [Mean (Standard Deviation); unit: units on a scale] — Subscale 1: How likely is it that in the next 3 months, you will refrain from smoking cigarettes...completely and permanently? when you get lonely? when you are with your friends who use them? when someone hands you a cigarette?
  Subscale 2: How likely is it that in the next 3 months, you will refrain from vaping nicotine...completely and permanently? when you get lonely? when you are with your friends who use them? when someone hands you a vape?
  Subscale items were summed & averaged; final scores ranged from 1 (worse outcome) to 4 (better outcome).
  units on a scale
    Subscale 1: Behavioral intentions to avoid cigarettes | 2.61 (0.81) | 2.49 (0.85) | 2.55 (0.83)
    Subscale 2: Behavioral intentions to avoid nicotine vapes | 2.29 (0.77) | 2.17 (0.67) | 2.23 (0.72)

OUTCOME MEASURES:

1. Primary Outcome: Visual Attention - Dwell Time
Description: Visual attention measured by dwell time (milliseconds) on areas of interest (AOI; e.g., text, graphic) within a stimuli was assessed via eye-tracking for each message (n=8). Dwell times on AOIs were summed for all stimuli viewed by each participant and averaged. Scores represent total average dwell time on AOIs across stimuli.
Time Frame: During intervention on Day 1, on average 3 minutes
Population: Participants were included for analysis if they completed the eye-tracking experiment and were not missing dwell time data.
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 65 | 71
milliseconds
  Textual AOI: Threat | 1871.00 [1732.95 to 2009.06] | 1881.01 [1763.64 to 1998.38]
  Textual AOI: Efficacy | 1695.21 [1570.14 to 1820.27] | 1603.15 [1488.94 to 1717.35]
  Textual AOI: Quit Resources | 317.90 [251.71 to 384.09] | 338.23 [278.62 to 397.84]
  Image AOI: Central Image | 2771.12 [2612.55 to 2929.69] | 2692.30 [2532.00 to 2852.60]
  Image AOI: Logo | 80.75 [52.88 to 108.61] | 97.80 [67.13 to 128.47]

2. Primary Outcome: Visual Attention - Time to First Fixation
Description: Time (milliseconds) to first fixation on areas of interest (text, graphic) within a stimuli was assessed via eye-tracking for each message (n=8). Time to first fixation on a specific AOI was summed for all stimuli viewed by each participant and averaged. Scores represent total average time to first fixation on AOIs across stimuli.
Time Frame: During intervention on Day 1, on average 3 minutes.
Population: Participants were included for analysis if they completed eye-tracking and did not have missing data capturing time to first fixation.
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 65 | 71
milliseconds
  Textual AOI: Threat | 890.45 [782.41 to 998.48] | 929.25 [826.81 to 1031.69]
  Textual AOI: Efficacy | 3525.47 [3320.72 to 3730.23] | 3494.96 [3303.00 to 3686.93]
  Textual AOI: Quit Resources | 1919.12 [1653.19 to 2185.06] | 1997.02 [1737.94 to 2256.10]
  Image AOI: Central Image | 1570.31 [1376.93 to 1763.70] | 1520.20 [1323.22 to 1717.18]
  Image AOI: Logo | 993.50 [775.40 to 1211.60] | 1061.08 [841.73 to 1280.42]

3. Primary Outcome: Perceived Message Effectiveness - Message Perceptions
Description: 6-items on a 5-point scale where 1 = Not at all and 5 = Very much.
  Please rate each statement from 1 (not at all) to 5 (very much). These message are worth remembering. These messages grabbed my attention. These messages are powerful. These messages are convincing. These messages are meaningful. These messages are informative.
  Individual items are summed and averaged for a total score ranging from 1 to 5. Higher scores indicate a better outcome.
Time Frame: Immediately post-exposure to intervention
Population: Analytic sample includes all participants for whom baseline and post-exposure data is available.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 83 | 82
score on a scale | 3.68 [3.46 to 3.90] | 3.7 [3.50 to 3.92]

4. Primary Outcome: Perceived Message Effectiveness - Effects Perceptions
Description: 6-items. 5-point scale where 1 = Strongly disagree to 5 = Strongly agree
  These messages discourage me from smoking cigarettes. These messages make me concerned about the negative effects of smoking cigarettes These messages make smoking cigarettes seem unpleasant to me.
  3-items above are summed and averaged. Higher scores indicate better outcome.
  These messages discourage me from vaping nicotine. These messages make me concerned about the negative effects of vaping nicotine. These messages make vaping nicotine seem unpleasant to me.
  3-items above are summed and averaged for a total score ranging from 1 to 5. Higher scores indicate a better outcome.
Time Frame: Immediately post-exposure to intervention
Population: Analytic sample includes all participants for whom baseline and post-exposure data is available.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 83 | 82
score on a scale
  Effects Perceptions: Smoking Cigarettes | 3.64 [3.44 to 3.84] | 3.80 [3.57 to 4.02]
  Effects Perceptions: Vaping Nicotine | 3.49 [3.27 to 3.72] | 3.69 [3.46 to 3.92]

5. Primary Outcome: Change in Behavioral Intentions
Description: 8 items total. 4-point scale 1 = Definitely not to 4 = Definitely will.
  The following items were asked at baseline and post-exposure.
  How likely is it that in the next 3 months, you will refrain from vaping nicotine....
  * completely and permanently?
  * when you get lonely?
  * when you are with your friends who use them?
  * when someone hands you a vape?
  How likely is it that in the next 3 months, you will refrain from smoking cigarettes...
  * completely and permanently?
  * when you get lonely?
  * when you are with your friends who use them?
  * when someone hands you a cigarette?
  For each subscale, pre-test and post-test items were summed and averaged. Change scores were calculated for each subscale by subtracting pre-test scores from post-test scores. Change scores could range from 0 to 3.
  Higher change scores indicate a better outcome (i.e. greater change in intentions to refrain from smoking or vaping)
Time Frame: Change from Baseline in behavioral intentions immediately post-exposure to intervention
Population: Analytic sample includes all participants for whom baseline and post-exposure data is available.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 83 | 82
score on a scale
  Change in cigarette smoking behavioral intentions | .20 [.05 to .35] | .36 [.21 to .51]
  Change in nicotine vaping behavioral intentions | .44 [.28 to .61] | .30 [.17 to .44]

6. Primary Outcome: Behavioral Intentions: Quitting Smoking
Description: Number of participants who answer "Yes" to the following: Do you plan to quit smoking cigarettes in the next 30 days? (Yes/No)
Time Frame: Difference between conditions in behavioral intentions to quit smoking at 1-week follow-up after intervention exposure
Population: Participants who reported current cigarette smoking at 1-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 35 | 33
Participants | 22 | 25

7. Primary Outcome: Behavioral Intentions to Quit Vaping
Description: Number of participants who answer "Yes" to the following: "Do you plan to quit vaping nicotine in the next 30 days?" (Yes/No)
Time Frame: Difference between conditions in behavioral intentions to quit vaping at 1-week follow-up after intervention exposure
Population: Participants reporting nicotine vaping at follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 39 | 39
Participants | 29 | 31

8. Secondary Outcome: Reactance
Description: 3-items; 5-point Likert scale where 1 = Strongly disagree and 5 = Strongly agree
  These messages are trying to manipulate me. These messages annoy me. The health effects of these messages are overblown.
  Items are summed and averaged for a total score ranging from 1 to 5. Higher scores indicate a worse outcome.
Time Frame: Immediately post-exposure to intervention
Population: Analysis includes all participants for whom baseline and post-exposure data is available.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 83 | 82
score on a scale | 2.11 [1.92 to 2.30] | 2.07 [1.86 to 2.29]

9. Secondary Outcome: Ad Relevance
Description: 5 items; 7-point Likert scale where 1 = Strongly Disagree and 7 = Strongly agree These ads were created just for me. These ads were created for people like me. These ads were relevant to me. These ads were of value to me. These ads were important to me.
  Items were summed and averaged for a total score ranging from 1 to 7. Higher scores indicate a better outcome.
Time Frame: Immediately post-exposure to intervention
Population: Analysis includes all participants for whom baseline and post-exposure data is available.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 83 | 82
score on a scale | 3.65 [3.39 to 3.91] | 3.64 [3.33 to 3.94]

10. Secondary Outcome: Liking
Description: Single item; 5-point Likert scale where 1 = Strongly disagree and 5 = Strongly agree
  I like these messages.
Time Frame: Immediately post-exposure to intervention
Population: Analysis includes all participants for whom baseline and post-exposure data is available.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 83 | 82
score on a scale | 3.82 [3.61 to 4.03] | 4.04 [3.81 to 4.26]

11. Secondary Outcome: Attitudes
Description: Two items; 7-point Likert scale where 1 = These message made me feel much worse and 7 = These message made me feel much better.
  Did these messages change how you feel about smoking combustible cigarettes?
  Did these messages change how you feel about vaping nicotine?
  Higher scores mean a worse outcome.
Time Frame: Immediately post-exposure to intervention
Population: Analysis includes all participants for whom baseline and post-exposure data is available.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 83 | 82
score on a scale
  Change in feelings about smoking cigarettes | 2.78 [2.49 to 3.07] | 2.94 [2.63 to 3.25]
  Change in feelings about vaping nicotine | 2.81 [2.52 to 3.09] | 2.90 [2.59 to 3.21]

12. Secondary Outcome: Response Efficacy
Description: 6-items; 5 point Likert scale where 1 = Strongly disagree and 5 = Strongly agree
  These messages will motivate CIGARETTE SMOKERS to switch to vaping. These messages will motivate people to quit ALL smoking and vaping. These messages will motivate NON-USERS to start vaping. These messages will motivate NON-USERS to start smoking cigarettes. These messages will motivate CIGARETTE SMOKERS to quit. These messages will motivate VAPERS to quit.
  Higher scores mean a better outcome.
Time Frame: Immediately post-exposure to intervention
Population: Analysis includes all participants for whom baseline and post-exposure data is available.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 83 | 82
score on a scale
  These messages will motivate CIGARETTE SMOKERS to switch to vaping. | 2.07 [1.82 to 2.33] | 1.93 [1.68 to 2.17]
  These messages will motivate people to quit ALL smoking and vaping. | 3.48 [3.23 to 3.73] | 3.43 [3.16 to 3.69]
  These messages will motivate NON-USERS to start vaping. | 1.53 [1.29 to 1.77] | 1.51 [1.29 to 1.74]
  These messages will motivate NON-USERS to start smoking cigarettes. | 1.46 [1.26 to 1.66] | 1.38 [1.20 to 1.55]
  These messages will motivate CIGARETTE SMOKERS to quit. | 3.41 [3.16 to 3.66] | 3.46 [3.20 to 3.73]
  These messages will motivate VAPERS to quit. | 3.34 [3.07 to 3.61] | 3.51 [3.26 to 3.76]

13. Secondary Outcome: Qualitative Recall of Health Messages
Description: Participants will be asked the following question: "The images that you viewed included health messages. What do you remember about the health messages?" Outcome indicates then number of participants who qualitatively reported recalling something about the health message.
Time Frame: 1-week follow-up after intervention exposure
Population: Number of participants who reported recalling something about the health messages.
Measure: Count of Participants; unit: Participants
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
Number analyzed (Participants) | 83 | 82
Participants | 81 | 79

ADVERSE EVENTS:
Time Frame: One week
Arm/Group | Culturally Targeted Messages | Non-targeted Messages
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/122
Other Adverse Events (participants affected / at risk) | 0/129 | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT05972941/Prot_SAP_000.pdf